CLINICAL TRIAL: NCT05864898
Title: Predictors of Failure of Non-invasive Ventilation and High Flow Nasal Cannula in Acute Respiratory Failure Patients : the Standardized PaO2 / FiO2 Ratio (P /F-st), ROX Index and HACOR
Brief Title: Predictors of Failure of Non-invasive Ventilation and High Flow Nasal Cannula
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hussein Makarem, Resident doctor, Assiut University
Other Study IDs: NIV and HFNC
Record Dates: First submitted 2023-03-22; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Acute Respiratory Failure Patients on NIV and HFNC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Comparison between some predictors of failure of non-invasive ventilation and high flow nasal cannula.

DETAILED DESCRIPTION:
Delayed intubation after NIV / HFNC failure is associated with high mortality rate in acute respiratory failure patients.

There are Many factors to predict early failure but World still searching for new factors and comparing between each ;in order to eatablish best one that achieve the least mortality rate.

Little studies about effiecacy of HACOR Score as a predictor of failure in HFNC patients.

Little studies about effiecacy of ROX Index as a predictor of failure in NIV ventilating patients.

ELIGIBILITY:
Inclusion Criteria:

Acute respiratory failure patients who need ventilatory Support either NIV or HFNC due to :

1. RR > 25 cycle / min
2. using accessory muscles and paradoxical breath.
3. PaO2 / FiO2 ratio < 300

Exclusion Criteria:

1. Absolute indication for intubation like coma, haemodynamically unstable… etc
2. Contr-indication of NIV like untreated Pneumothorax.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient in chest and Tuberculosis Departement, Assiut University
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Determine Golden time for intubation | 1 year
  Determine best time for intubation according to some predictors of failure of NIV and HFNC